CLINICAL TRIAL: NCT05237219
Title: The Effect of HEAT Therapy on patiEnts With Type 2 Diabetes Mellitus (HEATED): Protocol of a Randomized, Two-arm Controlled Trial
Brief Title: Heat Therapy in Patients With Type 2 Diabetes Mellitus
Acronym: HEATED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The human resources required to start enrollment were not available anymore.
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dr Hegyi Péter, Principal Investigator, Director of the Centre for Translational Medicine at University of Pécs, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 818-2/2022/EÜIG
Record Dates: First submitted 2022-01-05; First posted 2022-02-14 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: insulin resistance; balneotherapy; additional therapy; alternative therapy; heat shock proteins
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive heating (Experimental): Patients will be randomized to receive whole-body passive heating via 38°C natural thermal mineral water baths.
  Interventions: Procedure: Passive heating
- Thermoneutral (Active Comparator): Patients randomized to the comparator group will dip in thermoneutral natural thermal mineral water (30-32°C).
  Interventions: Procedure: Thermoneutral

INTERVENTIONS:
Procedure: Passive heating — Patients will perform baths in 38°C natural thermal mineral water a maximum of five times per week, over a 12-week period. This will result in a maximum of 60 visits. Each visit will take a maximum of 30 minutes with a physical check-up before and after the bath.
  Arms: Passive heating
Procedure: Thermoneutral — Patients will perform baths in 30-32°C natural thermal mineral water a maximum of five times per week, over a 12-week period. This will result in a maximum of 60 visits. Each visit will take a maximum of 30 minutes with a physical check-up before and after the bath.
  Arms: Thermoneutral

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a significant burden worldwide. In addition to lifestyle intervention, heat therapy has been shown to be effective in improving glycemic control. To date, there are no randomized, controlled trials investigating the efficacy of heat therapy in T2DM. Our aim is to investigate whether heat therapy with natural mineral water can improve blood glucose status in T2DM patients.

The HEATED study is a two-arm, randomized, controlled study. Patients with T2DM were randomly assigned to Group A (bath in 38 ° C natural thermal mineral water) or Group B (bath in thermoneutral water - 30-32 ° C). Both groups participate in up to five interventions per week, representing 50 to 60 heat therapies over the 12-week study. Each intervention lasts 30 minutes, preceded by a medical examination.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a significant burden worldwide. In addition to lifestyle intervention, heat therapy has been shown to be effective in improving glycemic control. To date, there are no randomized, controlled trials investigating the efficacy of heat therapy in T2DM. The study aims to investigate whether heat therapy with natural mineral water can improve blood glucose status in T2DM patients.

The HEATED study is a two-arm, randomized, controlled study. Patients with T2DM will be randomly assigned to Group A (bath in 38 ° C natural thermal mineral water) or Group B (bath in thermoneutral water - 30-32 ° C). Both groups will participate in up to five interventions per week, representing 50 to 60 heat therapies over the 12-week study. Each intervention will last 30 minutes, preceded by a medical examination. At baseline, patients' T2DM status will be recorded and possible micro- and macrovascular complications of T2DM are assessed by physical and laboratory tests. In addition, sensory and autonomic neuropathy will be assessed using Neurometer, Neuropad, and 128 Hz tuning fork tests. Quality of life will be assessed using the SF-36 questionnaire. In addition to baseline, patient data will be recorded at 4, 8, and 12 weeks. During routine blood collection, biobank storage will be performed via plus blood samples collection.

The primary endpoint will be the change from baseline in glycated hemoglobin by week 12 in both groups. Based on a preliminary estimate of the number of items, 65 patients per group are planned to be included in the HEATED study.

The results of the study described above may provide information on the utility of heat therapy in type 2 diabetics. Using the samples stored in the biobank, further analyzes will be performed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* patient with type 2 diabetes diagnosed according to the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD) guidelines
* serum glycated hemoglobin (HbA1c) level between 7 and 10% (53-86 mmol/mol)
* signed written informed consent form

Exclusion Criteria:

* other types of diabetes mellitus
* patients with poor glycaemic control or unstable diabetes
* patients with known serious comorbidity and/ or with advanced macrovascular complications
* active bacterial infection or treatment with antibiotics within 3 weeks
* open wounds or skin lesions
* history of skin-related conditions or sensitivity to prolonged water immersion or exposure to pool chemicals
* severe psychiatric pathology or psychosis
* pregnancy or breastfeeding
* judgment by medical provider that heat therapy/ hydrotherapy poses an undue burden or risk
* participating in other ongoing clinical trials
* heat or balneotherapy in the past 3 months
* morbid obesity (body mass index > 40 kg/m2)
* steroid treatment
* active autoimmune diseases
* coronavirus disease 2019 (COVID-19) in the past 3 months

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin A1c level | 12 weeks
  The absolut changes in the hemoglobin A1c from baseline to 12-weeks between the two groups will be compared.

SECONDARY OUTCOMES:
Change in hemoglobin A1c level | 4 and 8 weeks
  Absolute change from baseline to follow-up in hemoglobin A1c level.
Change in fasting plasma glucose | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in fasting plasma glucose.
Change in fasting insulin | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in fasting insulin.
Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).
Decrease of daily insulin dose | 4,8, and 12-weeks
  Absolute change from baseline to follow-up of the daily insulin dose.
Change in body mass index | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in body mass index. Weight and height will be combined to report BMI in kg/m^2.
Change in mean blood pressure | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in mean blood pressure.
Change in heart output | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in heart output.
Change in the prevalence of electrocardiogram events | 4,8, and 12-weeks
  Change in the prevalence of electrocardiogram events from baseline to follow-up. Electrocardiogram events represent a composite endpoint of any new events detected using a 12 lead electrocardiogram (e.g., myocardial infarction, atrial fibrillation, atrioventricular block, etc.).
Change in the proportion of hypertension | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in the proportion of hypertension
Change in the proportion of retinopathy | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in the proportion of retinopathy
Change in the proportion of nephropathy | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in the proportion of nephropathy
Change in the proportion of neuropathy | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in the proportion of neuropathy
Change in total cholesterol level | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in total cholesterol level.
Change in low-density lipoprotein cholesterol level | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in low-density lipoprotein cholesterol level.
Change in high-density lipoprotein cholesterol level | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in high-density lipoprotein cholesterol level.
Change in triglyceride level | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in triglyceride level.
Change in alkaline phosphatase (ALP) | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in alkaline phosphatase (ALP).
Change in alanine transaminase (ALT) | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in alanine transaminase (ALT).
Change in aspartate transaminase (AST) | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in aspartate transaminase (AST).
Change in gamma-glutamyl transferase (GGT). | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in gamma-glutamyl transferase (GGT).
Change in glomerular filtration rate | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in glomerular filtration rate.
Change in creatinine level | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in creatinine.
Change in thrombocyte aggregation | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in thrombocyte aggregation.
Heat Shock Protein expression | 4,8, and 12-weeks
  Difference between the two groups in the level of protein expression using flow cytometry.
Insulin signaling in polymorphonuclear cells | 4,8, and 12-weeks
  Difference between the two groups in the level of protein expression using flow cytometry.
Lipidom of polymorphonuclear cells | 4,8, and 12-weeks
  High sensitivity shotgun mass spectrometry will be used to characterize the lipidome of plasma, and polymorphonuclear blood cells.
Lipidom of plasma cells | 4,8, and 12-weeks
  High sensitivity shotgun mass spectrometry will be used to characterize the lipidome of plasma, and polymorphonuclear blood cells.
Change in obstructive sleep apnea proportion | 4,8, and 12-weeks
  Change in the proportion of obstructive sleep apnea from baseline to follow-up
Change in the proportion of abnormal overnight pulse oximetry | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in the proportion of abnormal overnight pulse oximetry.
Change in 24-hour blood pressure | 4,8, and 12-weeks
  Absolute change from baseline to follow-up in 24-hour blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Translational Medicine, University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sebok J, Edel Z, Vancsa S, Farkas N, Kiss S, Eross B, Torok Z, Balogh G, Balogi Z, Nagy R, Hooper PL, Geiger PC, Wittmann I, Vigh L, Dembrovszky F, Hegyi P. Heat therapy shows benefit in patients with type 2 diabetes mellitus: a systematic review and meta-analysis. Int J Hyperthermia. 2021;38(1):1650-1659. doi: 10.1080/02656736.2021.2003445. PMID 34808071
- [Background] Romeo GR, Lee J, Shoelson SE. Metabolic syndrome, insulin resistance, and roles of inflammation--mechanisms and therapeutic targets. Arterioscler Thromb Vasc Biol. 2012 Aug;32(8):1771-6. doi: 10.1161/ATVBAHA.111.241869. PMID 22815343
- [Background] Salas-Salvado J, Diaz-Lopez A, Ruiz-Canela M, Basora J, Fito M, Corella D, Serra-Majem L, Warnberg J, Romaguera D, Estruch R, Vidal J, Martinez JA, Aros F, Vazquez C, Ros E, Vioque J, Lopez-Miranda J, Bueno-Cavanillas A, Tur JA, Tinahones FJ, Martin V, Lapetra J, Pinto X, Daimiel L, Delgado-Rodriguez M, Matia P, Gomez-Gracia E, Diez-Espino J, Babio N, Castaner O, Sorli JV, Fiol M, Zulet MA, Bullo M, Goday A, Martinez-Gonzalez MA; PREDIMED-Plus investigators. Effect of a Lifestyle Intervention Program With Energy-Restricted Mediterranean Diet and Exercise on Weight Loss and Cardiovascular Risk Factors: One-Year Results of the PREDIMED-Plus Trial. Diabetes Care. 2019 May;42(5):777-788. doi: 10.2337/dc18-0836. Epub 2018 Nov 2. PMID 30389673
- [Background] Brunt VE, Howard MJ, Francisco MA, Ely BR, Minson CT. Passive heat therapy improves endothelial function, arterial stiffness and blood pressure in sedentary humans. J Physiol. 2016 Sep 15;594(18):5329-42. doi: 10.1113/JP272453. Epub 2016 Jun 30. PMID 27270841
- [Background] Hoekstra SP, Bishop NC, Faulkner SH, Bailey SJ, Leicht CA. Acute and chronic effects of hot water immersion on inflammation and metabolism in sedentary, overweight adults. J Appl Physiol (1985). 2018 Dec 1;125(6):2008-2018. doi: 10.1152/japplphysiol.00407.2018. Epub 2018 Oct 18. PMID 30335579
- [Background] Hooper PL, Balogh G, Rivas E, Kavanagh K, Vigh L. The importance of the cellular stress response in the pathogenesis and treatment of type 2 diabetes. Cell Stress Chaperones. 2014 Jul;19(4):447-64. doi: 10.1007/s12192-014-0493-8. Epub 2014 Feb 13. PMID 24523032
- [Background] Hooper PL. Hot-tub therapy for type 2 diabetes mellitus. N Engl J Med. 1999 Sep 16;341(12):924-5. doi: 10.1056/NEJM199909163411216. No abstract available. PMID 10498473
- [Derived] Sebok J, Edel Z, Dembrovszky F, Farkas N, Torok Z, Balogh G, Peter M, Papp I, Balogi Z, Nusser N, Peter I, Hooper P, Geiger P, Eross B, Wittmann I, Vancsa S, Vigh L, Hegyi P. Effect of HEAT therapy in patiEnts with type 2 Diabetes mellitus (HEATED): protocol for a randomised controlled trial. BMJ Open. 2022 Jul 12;12(7):e062122. doi: 10.1136/bmjopen-2022-062122. PMID 35820741
- See also: Related info — https://tm-centre.org/en/research/clinical-trials/